CLINICAL TRIAL: NCT05006144
Title: Effects of Selective Dorsal Rhizotomy on Trunk Control, Selectivity and Upper Extremity Function of Non-ambulant Children With Bilateral Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Effects of Selective Dorsal Rhizotomy on Non-ambulant Children With Bilateral Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physiacl therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: spastic cerebral palsy
Record Dates: First submitted 2021-08-07; First posted 2021-08-16 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Bilateral Cerebral Palsy
Keywords: Bilateral Cerebral Palsy; Selective dorsal rhizotomy; segmental trunk control; Motor development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Random allocation of participants will be completed using a random number generator, with the allocation to either the control or selective dorsal rhizotomy group being concealed. The random numbers are generated by the principle physical therapists with every alternate number being marked either "1" or "2." However, the receptionist was blinded to the interventions assigned to group 1 (control group) and group 2 (SDR group). During allocation, every parent/legal guardian is asked to pick up one enclosed envelope from a box containing numbers from 1 to 30. Then, they are allocated to either group 1 or group 2 to minimize the risk of allocation bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): control group
  Interventions: Other: sequenced trunk co-activation exercises; Other: Standard Orthotic Management
- Experimental group (Experimental): selective dorsal rhizotomy
  Interventions: Other: sequenced trunk co-activation exercises; Other: Standard Orthotic Management; Other: selective dorsal rhizotomy

INTERVENTIONS:
Other: sequenced trunk co-activation exercises — * Sequenced trunk co-activation exercises were basically used for facilitation of functional activities through trunk musculature dynamic co-activation of in the lateral plane which is required for basic developmental milestones. In the frontal plane, encourage the child to actively shift his/her weight to maintain the weight-bearing side straight while keeping proper active co-activation of trunk musculature. Efficient trunk rotation is essential for acquiring of equilibrium reactions and balance. Enhancement of efficient active trunk rotation as the child could achieve active trunk musculature co-activation while maintaining the weight-bearing side straight (Arndt et al., 2008).
  * Righting and protective reactions
  * Functional stretching exercises.
Other: Standard Orthotic Management — A custom-made articulating ankle foot orthosis with a hinge at the level of the medial malleolus of the ankle is fabricated for each child from the same copolymer thermoplastic mold after casting with the subtalar joint in neutral position. The orthosis extended distally to the tip of the toes and proximally on the posterior surface of the leg to about 5 cm below the knee and secured to the foot by three straps across the forefoot, the front of the ankle, and to the anterior upper tibial portion. It is fabricated to permit free ankle dorsiflexion and lock the plantar flexion at 0 dorsiflexion. The splinting schedule started gradually for 2 h/day in the first month, 4 h/day in the second month to the entire wake-up time of the day in the third and fourth months to accommodate children to the orthosis.
Other: selective dorsal rhizotomy — All SDRs were performed by a single neurosurgeon through an osteoplastic laminotomy from L2 to L5 that left the facet joints intact. After opening the dura, the posterior nerve roots of L2 to S1 were identified and divided into 3 to 6 rootlets. At L2, from 30% to 50% of the posterior nerve rootlets were sectioned without selective stimulation. Selective electric stimulation of each nerve rootlet was performed from L3 to S1. The percentage of rootlets sectioned at each level (table 3) was determined by the surgical team based on the electromyographic results obtained intrasurgically and knowledge of the presurgical assessment results. The laminae were replaced on the completion of the rootlet stimulation and secured with sutures in the yellow ligament and the supraspinous ligament.
  Arms: Experimental group

SUMMARY:
Children with spastic bilateral cerebral palsy are late developers. delayed gross and fine motor development require early intervention to improve the child performance and avoid secondary impairments.

DETAILED DESCRIPTION:
increased tone of lower extremity muscles interfere with the child sitting posture and trunk control. delayed sitting and lack of trunk control contribute to the impairments of upper extremity functions.

selective dorsal rhizotomy is a surgical procedure to control increased tone of the lower extremities. Therefore, the current study is carried out to investigate the effects of selective dorsal rhizotomy on trunk control, selectivity and upper extremity function of non-ambulant children with bilateral spastic cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* CP, spastic diplegia
* 4-7 years of age
* On Level IV-V on Gross Motor Function Classification System
* At least six months after the last Botulinum toxin A injection in the lower extremities
* Average intelligent quotient according to medical records for active participation
* Partial trunk control (sitting with support).

Exclusion Criteria:

* Structural non-reducible deformities or musculoskeletal surgery in the lower extremities in the past 12 months
* Ankle clonus
* Exaggerated deep tendon reflex in the legs
* Babinski sign;
* Moderate to severe signs of dystonia, athetosis or ataxia.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Segmental trunk control | period of the treatment was 4 successive months
  The Segmental Assessment of Trunk Control is applied to assess upright trunk postural control in sitting position based on subdividing the trunk into 6 segments. The head/trunk control is acquired segment by segment if upright sitting posture can be maintained under three conditions including: static control at static position, active control while the child moves the head and/or arm and reactive control after external perturbation.The trunk segments according to the scale include: head/neck, thoracic (upper, mid and lower) and lumbar (upper and lower) segments. It is an ordinal scale with a grade 1 to 7 is assigned for each segment with the score 7 indicates that the infant can't retain independent sitting (no hand support). A score of 8 is given as full trunk control is gained.
Gross motor function | period of the treatment was 4 successive months
  The gross motor function measure-88 is a valid and reliable criterion referenced instrument; is currently used to evaluate the motor function over time in individuals with cerebral palsy. It consists of 5 sections including; A) lying and rolling, B) sitting, C) crawling and kneeling, D) standing; E) walking, running, jumping. Each item was scored on a four-point scale as 0, 1, 2 or 3 with higher scores representing a better performance. The scoring key was; 0=does not initiate, 1=initiates the task (<10%), 2=partial completion of the task (10% to <100%), 3=task completed (100%). If an item was not tested it was marked as not tested

SECONDARY OUTCOMES:
upper extremity function | period of the treatment was 4 successive months
  The quality of upper extremity skill test is a reliable and valid tool used to measure the motor function in children with cerebral palsy ages of 18 months to 8 years. The assessment procedures were conducted according to the instruction manual to assess the movement patterns in four basic domains representing dissociated movement; grasp; protective extension; and weight bearing. The total scores for each domain percentage score are calculated as total score which range from zero to 100% with higher score reflects better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem A Aly, Phd, Study Chair — PhD of physical therapy for pediatrics, faculty of physical therapyCairo university; Ahmed rabie, Phd, Study Director — Department of neurosurgery, faculty of medicine , Alexandria university
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt